CLINICAL TRIAL: NCT03645759
Title: Improving Quality of Life for Veterans With Stroke and Psychological Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2898-P; I21RX002898-01A1 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Depression; Anxiety
Keywords: behavioral treatment; telehealth; stroke self-management; psychological distress; social integration
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Behavioral treatment intervention that focuses on enhancing stroke self-management, psychological distress and social functioning that will be provided to two groups (treatment and education plus usual care).
Who Masked: Participant, Investigator
Masking Description: No other parties will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I'm Whole (Experimental): This arm will receive 6 behavioral health treatment sessions that focus on stroke self-management, psychological distress and social re-integration. Treatments will occur weekly. They will also receive 3 assessments at 0, 6, and 12 weeks.
  Interventions: Behavioral: I'm Whole
- Education + usual care (Active Comparator): This arm will only receive the standard usual care for stroke self-management provided by the Michael E. Debakey VA Medical facility and will receive 6 brief health education calls unrelated to stroke or psychological distress.
  Interventions: Other: Education + usual care

INTERVENTIONS:
Behavioral: I'm Whole — I'm whole will provide 6 behavioral health treatment sessions that focus on stroke self-management, psychological distress and social re-integration.
  Arms: I'm Whole
Other: Education + usual care — Will receive the standard usual care for stroke self-management provided by the Michael E. Debakey VA Medical facility and will receive 6 brief health education calls unrelated to stroke or psychological distress.
  Arms: Education + usual care

SUMMARY:
The study will create a treatment to improves mobility, physical activity, engagement in activities with family and friends and overall satisfaction with life for Veterans who have depression and anxiety after having a stroke. The treatment will then be tested to ensure it makes the desired improvements in the Veterans.

DETAILED DESCRIPTION:
The study has three aims. The first aim is to develop a client-centered, behavioral stroke self-management program (I'm Whole) for Veterans with stroke and psychological distress (e.g., symptoms of anxiety and/or depression). This will be done using expert input from a multidisciplinary team of a clinical psychologist, nurse practitioner, exercise physiologist and social role functioning expert will be used to create the I'm Whole patient workbook and clinician manual.

The second aim is to pilot the I'm Whole treatment by delivering the intervention to 5 Veterans suffering from stroke and comorbid depression and/or anxiety symptoms. The feasibility (barriers and facilitators to completing I'm Whole and acceptability of the intervention) will be assessed through qualitative interviews posttreatment. Veterans' feedback about ways to improve I'm Whole will be analyzed and used to improve treatment.

The third aim is to test the feasibility and preliminary efficacy of I'm Whole on quality of life (primary outcome) physical functioning, physical activity, social role functioning, psychological distress, and satisfaction with I'm Whole (secondary outcomes). To test the feasibility and efficacy, a small randomized controlled trial (RCT) with 30 Veterans (15 I'm Whole and 15 education+usual care) with stroke and psychological distress will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* a documented history of stroke and/or transient ischemic attack within the last 30 days
* a modified Rankin score of > 3)
* regular access to a computer or tablet with internet and a camera
* ability to give appropriate informed consent
* score > 5 on a measure of depression (Patient Health Questionnaire [PHQ-8]) and/or >17 on a measure of anxiety (Generalized Anxiety Disorder-7 [GAD-7]) assessments
* ability to ambulate with or without assistance of a cane or walker

Exclusion Criteria:

* cognitive impairment, as evidenced by a score of >3 on a brief cognitive screener
* documented diagnosis of psychotic disorder or schizophrenia
* documented severe depression, anxiety (based on PHQ-8 or GAD-7 score of > 20), or hospitalization for psychiatric illness within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina L. Evans, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- I'm Whole: This arm will receive 6 behavioral health treatment sessions that focus on stroke self-management, psychological distress and social re-integration. Treatments will occur weekly. They will also receive 3 assessments at 0 and 12 weeks.
  I'm Whole: I'm whole will provide 6 behavioral health treatment sessions that focus on stroke self-management, psychological distress and social re-integration.
Period: Overall Study
Arm/Group | I'm Whole | Education + Usual Care
Started | 19 | 19
Completed | 16 | 17
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I'm Whole | Education + Usual Care | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.44 (3.77) | 63.44 (4.27) | 64.44 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 17 | 19 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 9 | 24
  White | 4 | 10 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 38
International physical activity questionnaire [Mean (Standard Deviation); unit: MET Minutes per day] | 203 (284) | 143 (233.9) | 173 (258.8)
Sedentary Behaviors Questionnaire [Mean (Standard Deviation); unit: hours spent in sedentary behaviors] | 5.73 (9.49) | 4.51 (1.40) | 5.12 (5.45)
Community Integration Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Total score range is 13-39. Lower values represent a better outcome and greater integration into the community.
  units on a scale | 18.60 (4.60) | 29.70 (4.41) | 24.15 (4.51)
Patient-Reported Outcomes Measurement Information System [Mean (Standard Deviation); unit: units on a scale] — The scores range from 0 - 100. Higher scores indicate greater difficulties with overall health functioning.
  units on a scale | 64.04 (5.32) | 61.01 (9.10) | 62.53 (7.21)
Generalized Anxiety Disorder-7 items [Mean (Standard Deviation); unit: units on a scale] — Total score range is 0-21. Lower values represent a better outcome and less symptoms of anxiety.
  units on a scale | 4.80 (0.70) | 4.52 (1.01) | 4.65 (0.85)
Patient Health Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Total score range is 0-24. Lower values represent a better outcome and less symptoms of depression.
  units on a scale | 11.01 (0.91) | 10.10 (0.70) | 10.55 (0.81)
36-Item Short Form Survey [Mean (Standard Deviation); unit: units on a scale] — 0 to 100, with lower scores denoting poorer health
  units on a scale | 40.23 (9.15) | 51.39 (10.96) | 45.81 (10.06)

OUTCOME MEASURES:

1. Primary Outcome: Stroke Specific Quality of Life Scale Change
Description: The Stroke Specific Quality of Life Scale assesses change in energy, language, vision, mobility, fine motor tasks, mood, personality and thinking, social roles, family roles and work productivity. Scores are reported for the energy, language, mobility, personality, mood, family roles, thinking, and social roles. The score range for each item 1= strongly disagree to 5=strongly agree with a higher score indicating greater disability and worst outcomes. A total score range is 14-70.
Time Frame: Absolute values at 12 weeks post-treatment are being reported
Population: Estimates of changes in patient-reported outcomes were calculated using intent to-treat approach. The paired change in outcome scores from baseline to the end of the study and differences in paired change in scores in treatment and EUC arms were compared with zero using Wilcoxon's signed-rank test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I'm Whole | Education + Usual Care
Number analyzed (Participants) | 16 | 17
units on a scale | 41.24 (6.30) | 41.67 (5.80)

2. Secondary Outcome: Physical Activity and Disability Survey Change
Description: The Physical Activity and Disability Survey measures change in exercise, leisure time physical activity, indoor and outdoor household activity, wheelchair ambulation, employment-related activity and rehabilitation therapy-related activity. Scores were reported for each 6 areas of exercise/activity. The subscale score is based on the self-reported amount of time an individual states they spend performing each exercise. Higher values represent a better outcome and more time spent engaging in the activity. The range of scores are 0-1440 minutes per day.
Time Frame: The absolute values at 12 weeks post-treatment are being reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I'm Whole | Education + Usual Care
Number analyzed (Participants) | 16 | 17
units on a scale | 602 (48) | 60 (22)

3. Secondary Outcome: Community Integration Questionnaire Change
Description: The Community Integration Questionnaire measures change in home integration (i.e., market, meal preparation, household activities, finance), social integration (i.e., shopping, avocation, going out), and productive activity (i.e., work, school, volunteer activity). The score range is 1=you yourself alone 3=someone else. Total score range is 13-39. Lower values represent a better outcome and greater integration into the community.
Time Frame: The absolute values at 12 weeks post-treatment are being reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I'm Whole | Education + Usual Care
Number analyzed (Participants) | 16 | 17
units on a scale | 16.8 (4.21) | 13.8 (4.23)

4. Secondary Outcome: Patient Health Questionnaire-8 Item Change
Description: The Patient Health Questionnaire-8 assesses change in severity of depression symptoms over the last two weeks. The score range is 0=Not at all to 3=Nearly every day. Total score range is 0-24. Lower values represent a better outcome and less symptoms of depression.
Time Frame: The absolute values at 12 weeks post-treatment are being reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I'm Whole | Education + Usual Care
Number analyzed (Participants) | 16 | 17
units on a scale | 4.00 (1.10) | 8.21 (0.80)

5. Secondary Outcome: General Anxiety Disorder-7 Change
Description: The General Anxiety Disorder-7 assesses change in severity of anxiety symptoms over the last two weeks. The total score is reported. The score range is 0=Not at all to 3=Nearly every day. Total score range is 0-21. Lower values represent a better outcome and less symptoms of anxiety.
Time Frame: The absolute values at 12 weeks post-treatment are being reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I'm Whole | Education + Usual Care
Number analyzed (Participants) | 16 | 17
units on a scale | 2.80 (0.82) | 3.91 (1.03)

ADVERSE EVENTS:
Time Frame: Adverse data was collected for 1 year and 6 months.
Description: The definition does not differ from that defined by clinicaltrials.gov.
Arm/Group | I'm Whole | Education + Usual Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
The small sample size is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03645759/Prot_SAP_000.pdf